CLINICAL TRIAL: NCT02827006
Title: CaP Cement is Equivalent to Iliac Bone Graft in Filling of Large Metaphyseal Defects: A 2 Year Prospective Randomised Study on Distal Radius Osteotomies
Brief Title: CaP Cement is Equivalent to Iliac Bone Graft in Filling of Large Metaphyseal Defects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Mona Winge, Consultant, Orthopaedic Surgeon, Principal Investigator, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06/8465
Record Dates: First submitted 2016-06-27; First posted 2016-07-11 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Dorsal Malunion of the Distal Radius
Keywords: Bone graft; Calcium phosphate bone cement; RCT; Xray; CT

STUDY DESIGN:
Intervention Model Description: the standard treatment is a corrective osteotomy with bone graft. The intervention in parallel group is a corrective osteotomy and use of CaP bone cement
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bone graft (Active Comparator): Bone graft from iliac crest as gapfiller
  Interventions: Procedure: corrective osteotomy distal radius
- Calcium phosphate bone cement (Experimental): CaP bone cement as gapfiller
  Interventions: Procedure: corrective osteotomy distal radius

INTERVENTIONS:
Procedure: corrective osteotomy distal radius — Opening wedge corrective osteotomy on dorsal malunions of the distal radius. Distraction and correction of deformity.

SUMMARY:
CaP Cement is Equivalent to Iliac Bone Graft in Filling of Large Metaphyseal Defects

DETAILED DESCRIPTION:
Background: A bone graft from the iliac crest has long been the gold standard for filling voids in opening wedge osteotomies. CaP bone cement has been considered the possible alternative to bone graft.

Methods: 20 adult patients with distal radius malunions and dorsal deformities were randomised intra-operatively to bone graft (10) or CaP bone cement (10). Dorsal titanium locking plates were used and the wrist was stabilised in a cast for 8 weeks. Follow-ups for 24 months included VAS on wrist and iliac crest, grip strength, ROM bilaterally, Quick-DASH and Gartland & Werley's functional scoring system. X-rays and CT scans were taken at 8 wks, 3-6-12-24 mths.

ELIGIBILITY:
Inclusion Criteria:

* distal radius malunion with dorsal deformity, disability and pain.

Exclusion Criteria:

* age under 18 years, bad health, inflammatory arthritis and radio-carpal osteoarthritis.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
volar angulation distal radius, x-ray | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Magne Røkkum, MD PhD, Study Director — OUS RH

IPD SHARING:
Plan to Share IPD: Yes